CLINICAL TRIAL: NCT00916357
Title: Phase 2, Double-Blind Randomized, 3-way Cross-Over Liquid Meal Study With Optimal Doses of SC Administered Insulin Lispro With and Without rHuPH20 and Regular Human Insulin With rHuPH20 to Compare Pharmacokinetics, Postprandial Glycemic Response, and Optimal Insulin Dose in Patients With T2DM
Brief Title: Liquid Meal Study With Insulin Lispro With/Without Recombinant Human Hyaluronidase PH20 (rHuPH20) and Regular Human Insulin With rHuPH20 to Compare Pharmacokinetics, Postprandial Glycemic Response, and Optimal Insulin Dose in Participants With Type 2 Diabetes Mellitus (T2DM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: HALO-117-204
Record Dates: First submitted 2009-06-05; First posted 2009-06-09 (Estimated); Results first posted 2014-08-18 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: recombinant human hyaluronidase PH20 (rHuPH20); Insulin lispro; Regular human insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Insulin Lispro; Insulin; Insulin, Regular, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Humalog, Then Humalog + rHuPH20, Then Humulin-R + rHuPH20 (Active Comparator): A subcutaneous (SC) injection of 0.3- to 0.5-units per kilogram (U/kg) of Humalog alone for up to 3 dose-finding (DF) visits (each visit separated by a 3- to 14-day washout period), followed by a SC injection of the appropriate dose of Humalog. After a 3- to 14-day washout period, the DF process and injection of appropriate dose was repeated with 0.3- to 0.5-U/kg Humalog + 3.75 nanograms/kilogram (ng/kg) recombinant human hyaluronidase PH20 (rHuPH20). The DF process and injection of appropriate dose was then repeated with 0.3- to 0.5-U/kg Humulin-R + 3.75 ng/kg rHuPH20 following a 3 to 14 day washout period.
  Interventions: Drug: Humalog; Drug: Humulin-R; Drug: Recombinant human hyaluronidase PH20 (rHuPH20)
- Humalog, Then Humulin-R + rHuPH20, Then Humalog + rHuPH20 (Active Comparator): A subcutaneous (SC) injection of up to 0.3- to 0.5-units per kilogram (U/kg) of Humalog alone for up to 3 dose finding (DF) visits (each visit separated by a 3- to 14-day washout), followed by a single SC injection of the appropriate dose of Humalog. After a 3- to 14-day washout period, the DF process and injection of appropriate dose was repeated with 0.3- to 0.5-U/kg Humulin-R + 3.75 nanograms/kilogram (ng/kg) recombinant human hyaluronidase PH20 (rHuPH20). The DF process and injection of appropriate dose was then repeated with 0.3- to 0.5-U/kg Humalog + 3.75 ng/kg rHuPH20 following a 3- to 14-day washout period.
  Interventions: Drug: Humalog; Drug: Humulin-R; Drug: Recombinant human hyaluronidase PH20 (rHuPH20)
- Humalog + rHuPH20, Then Humalog, Then Humulin-R + rHuPH20 (Active Comparator): A subcutaneous (SC) injection of up to 0.3- to 0.5-units per kilogram (U/kg) of Humalog + 3.75 nanograms per kilogram (ng/kg) recombinant human hyaluronidase PH20(rHuPH20) for up to 3 dose-finding (DF) visits (each visit separated by a 3- to 14-day washout), followed by a single SC injection of the appropriate dose of Humalog + rHuPH20. After a 3- to 14-day washout period, the DF process and injection of appropriate dose was repeated with 0.3- to 0.5-U/kg Humalog alone. The DF process and injection of appropriate dose was then repeated with 0.3- to 0.5-U/kg Humulin-R + 3.75 ng/kg rHuPH20 following a 3- to 14-day washout period.
  Interventions: Drug: Humalog; Drug: Humulin-R; Drug: Recombinant human hyaluronidase PH20 (rHuPH20)
- Humalog + rHuPH20, Then Humulin-R + rHuPH20, Then Humalog (Active Comparator): A subcutaneous (SC) injection of up to 0.3- to 0.5-units per kilogram (U/kg) of Humalog + 3.75 nanograms per kilogram (ng/kg) of recombinant human hyaluronidase PH20 (rHuPH20) for up to 3 dose finding (DF) visits (each visit separated by a 3- to 14-day washout), followed by a single SC injection of the appropriate dose of Humalog + rHuPH20. After a 3- to 14-day washout period, the DF process and injection of appropriate dose was repeated with 0.3- to 0.5-U/kg Humulin-R + rHuPH20. The DF process and injection of appropriate dose was then repeated with 0.3- to 0.5-U/kg Humalog following a 3- to 14-day washout period.
  Interventions: Drug: Humalog; Drug: Humulin-R; Drug: Recombinant human hyaluronidase PH20 (rHuPH20)
- Humulin-R + rHuPH20, Then Humalog, Then Humalog + rHuPH20 (Active Comparator): A subcutaneous (SC) injection of up to 0.3- to 0.5-units per kilogram (U/kg) of Humulin-R + 3.75 nanograms per kilogram (ng/kg) of recombinant human hyaluronidase PH20 (rHuPH20) for up to 3 dose-finding (DF) visits (each visit separated by a 3- to 14-day washout), followed by a single SC injection of the appropriate dose of Humulin-R + rHuPH20. After a 3- to 14-day washout period, the DF process and injection of appropriate dose was repeated with 0.3- to 0.5-U/kg Humalog alone. The DF process and injection of appropriate dose was then repeated with 0.3- to 0.5-U/kg Humalog + 3.75 ng/kg rHuPH20 following a 3- to 14-day washout period.
  Interventions: Drug: Humalog; Drug: Humulin-R; Drug: Recombinant human hyaluronidase PH20 (rHuPH20)
- Humulin-R + rHuPH20, Then Humalog + rHuPH20, Then Humalog (Active Comparator): A subcutaneous (SC) injection of 0.3- to 0.5-units per kilogram (U/kg) of Humulin-R + 3.75 nanograms per kilogram (ng/kg) of recombinant human hyaluronidase PH20 (rHuPH20) for up to 3 dose-finding (DF) visits (each visit separated by a 3- to 14-day washout), followed by a single SC injection of the appropriate dose of Humulin-R + rHuPH20. After a 3- to 14-day washout period, the DF process and injection of appropriate dose was repeated with 0.3- to 0.5-U/kg Humalog + 3.75 ng/kg rHuPH20. The DF process and injection of appropriate dose was then repeated with 0.3- to 0.5-U/kg Humalog alone following a 3- to 14-day washout period.
  Interventions: Drug: Humalog; Drug: Humulin-R; Drug: Recombinant human hyaluronidase PH20 (rHuPH20)

INTERVENTIONS:
Drug: Humalog
  Other Names: Insulin lispro
Drug: Humulin-R
  Other Names: Humulin; Regular human insulin
Drug: Recombinant human hyaluronidase PH20 (rHuPH20)
  Other Names: PH20; HYLENEX

SUMMARY:
This is a single-center, Phase 2, randomized, double-blind, 3-way crossover meal study in participants with Type 2 Diabetes Mellitus (T2DM) to determine the optimum dose and compare the pharmacokinetics (PK) and postprandial glycemic response of Humalog alone, Humalog + recombinant human hyaluronidase PH20 (rHuPH20), and Humulin-R + rHuPH20 administered subcutaneously.

DETAILED DESCRIPTION:
This study design was chosen to assess the differences between pharmacokinetic (PK) and pharmacodynamic (PD) parameters, including postprandial glycemic response, of Humalog + recombinant human hyaluronidase PH20 (rHuPH20), Humalog alone, and Humulin-R + rHuPH20 at optimal doses following a liquid meal.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of age 18 to 70 years, inclusive
* Participants with Type 2 diabetes mellitus (T2DM) per World Health Organization criteria treated with basal and/or bolus insulin for ≥12 months.
* Body mass index (BMI) between 18 to 45 kilograms per square meter (kg/m^2), inclusive
* Glycosylated hemoglobin A1c (HbA1c) ≤10%
* Current treatment with insulin ≥60 Units/day (U/d)
* A participant taking oral hypoglycemic agents must be on a stable dose for >8 weeks with the exception of thiazolidinediones (TZD), which should be >12 weeks.
* Total body weight >65 kilograms (kg) (143 pounds [lb]) for men and >46 kg (101 lb) for women
* Vital signs (blood pressure [BP], pulse rate, and body temperature) within normal range or, if out of range, assessed by the Investigator as not clinically significant (NCS)
* Participants should be in good general health based on medical history and physical examination without medical conditions that might prevent the completion of study drug injections and assessments in this protocol
* Decision making capacity and willingness to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures including adequate venous access.
* Signed and written Internal Review Board-approved informed consent

Exclusion Criteria:

* Known or suspected allergy to any components of any of the study drugs in this study
* Previous enrollment in this study
* A participant who has proliferative retinopathy, proliferative maculopathy, and/or severe neuropathy (in particular, autonomic neuropathy) as judged by the Investigator
* As judged by the Investigator, clinically significant active disease of the gastrointestinal, cardiovascular (including a history of arrhythmia or conduction delays on electrocardiogram [ECG] and New York Heart Association [NYHA] Class III/IV heart disease), hepatic, neurological, renal, genitourinary, or hematological systems
* As judged by the Investigator, uncontrolled hypertension (diastolic BP ≥100 millimeters of mercury [mmHg] and/or systolic BP ≥160 mmHg after 5 minutes in the supine position).
* As judged by the Investigator, clinically significant findings in routine laboratory data (anemia with hematocrit less than 33% at screening is specifically exclusionary)
* Positive human immunodeficiency virus (HIV) antibody test, hepatitis B (anti-HBsAg), or hepatitis C (anti-HCV) antibody test
* Current addiction to alcohol or substances of abuse as determined by the Investigator
* Known use of drugs (other than oral hypoglycemic agents) that may interfere with the interpretation of study results or are known to cause clinically relevant interference with insulin action, glucose utilization, or recovery from hypoglycemia
* Recurrent major hypoglycemia or hypoglycemic unawareness as determined by the Investigator
* Mental incapacity, unwillingness, or language barriers precluding adequate understanding or cooperation in this study
* Symptomatic gastroparesis
* Donation of blood in excess of 500 milliliters (mL) within 56 days before dosing
* Use of any investigational drug or device 30 days before enrollment in this study
* Pregnancy, breast-feeding, the intention of becoming pregnant, or not using adequate contraceptive measures (adequate contraceptive measures consist of sterilization, intra-uterine device [IUD], oral or injectable contraceptives, barrier methods, or remaining abstinent)
* Any condition (intrinsic or extrinsic) that, in the judgment of the Investigator, will interfere with study participation or evaluation of data

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-07; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Hompesch, M.D., Principal Investigator — Profil Institute for Clinical Research, Inc.
Locations (1):
- Profil Institute for Clinical Research, Inc., Chula Vista, California, United States

REFERENCES:
- [Result] Hompesch M, Muchmore DB, Morrow L, Ludington E, Vaughn DE. Improved postprandial glycemic control in patients with type 2 diabetes from subcutaneous injection of insulin lispro with hyaluronidase. Diabetes Technol Ther. 2012 Mar;14(3):218-24. doi: 10.1089/dia.2011.0117. Epub 2011 Dec 2. PMID 22136324

RESULTS

PARTICIPANT FLOW:
Groups:
- Humalog, Then Humalog + rHuPH20, Then Humulin-R + rHuPH20: A subcutaneous (SC) injection of up to 0.3- to 0.5-units per kilogram (U/kg) of Humalog alone for up to 3 dose-finding (DF) visits (each visit separated by a 3- to 14-day washout period), followed by a SC injection of the appropriate dose of Humalog. After a 3- to 14-day washout period, the DF process and injection of appropriate dose was repeated with up to 0.3- to 0.5-U/kg Humalog + 3.75 nanograms/kilogram (ng/kg) recombinant human hyaluronidase PH20 (rHuPH20). The DF process and injection of appropriate dose was then repeated with 0.3- to 0.5-U/kg Humulin-R + 3.75 ng/kg rHuPH20 following a 3- to 14-day washout period.
- Humalog + rHuPH20, Then Humalog, Then Humulin-R + rHuPH20: A subcutaneous (SC) injection of up to 0.3- to 0.5-units per kilogram (U/kg) of Humalog + 3.75 nanograms per kilogram (ng/kg) recombinant human hyaluronidase PH20 (rHuPH20) for up to 3 dose-finding (DF) visits (each visit separated by a 3- to 14-day washout), followed by a single SC injection of the appropriate dose of Humalog + rHuPH20. After a 3- to 14-day washout period, the DF process and injection of appropriate dose was repeated with 0.3- to 0.5-U/kg Humalog alone. The DF process and injection of appropriate dose was then repeated with 0.3- to 0.5-U/kg Humulin-R + 3.75 ng/kg rHuPH20 following a 3- to 14-day washout period
- Humulin-R + rHuPH20, Then Humalog, Then Humalog + rHuPH20: A subcutaneous (SC) injection of up to 0.3- to 0.5-units per kilogram (U/kg) of Humulin-R + 3.75 nanograms per kilogram (ng/kg) of recombinant human hyaluronidase PH20 (rHuPH20) for up to 3 dose-finding (DF) visits (each visit separated by a 3- to 14-day washout), followed by a single SC injection of the appropriate dose of Humulin-R + rHuPH20. After a 3- to 14-day washout period, the DF process and injection of appropriate dose was repeated with 0.3- to 0.5-U/kg Humalog alone. The DF process and injection of appropriate dose was then repeated with 0.3-to 0.5-U/kg Humalog + 3.75 ng/kg rHuPH20 following a 3- to 14-day washout period.
- Humulin-R + rHuPH20, Then Humalog + rHuPH20, Then Humalog: A subcutaneous (SC) injection of up to 0.3- to 0.5-units per kilogram (U/kg) of Humulin-R + 3.75 nanograms per kilogram (ng/kg) of recombinant human hyaluronidase PH20 (rHuPH20) for up to 3 dose-finding (DF) visits (each visit separated by a 3- to 14-day washout), followed by a single SC injection of the appropriate dose of Humulin-R + rHuPH20. After a 3- to 14-day washout period, the DF process and injection of appropriate dose was repeated with 0.3- to 0.5-U/kg Humalog + 3.75 ng/kg rHuPH20. The DF process and injection of appropriate dose was then repeated with 0.3- to 0.5-U/kg Humalog alone following a 3- to 14-day washout period.
Period: Period 1
Arm/Group | Humalog, Then Humalog + rHuPH20, Then Humulin-R + rHuPH20 | Humalog, Then Humulin-R + rHuPH20, Then Humalog + rHuPH20 | Humalog + rHuPH20, Then Humalog, Then Humulin-R + rHuPH20 | Humalog + rHuPH20, Then Humulin-R + rHuPH20, Then Humalog | Humulin-R + rHuPH20, Then Humalog, Then Humalog + rHuPH20 | Humulin-R + rHuPH20, Then Humalog + rHuPH20, Then Humalog
Started | 4 | 4 | 4 | 4 | 3 | 4
Received at Least 1 Dose of Study Drug | 4 | 4 | 4 | 4 | 3 | 4
Completed | 3 | 4 | 4 | 4 | 3 | 4
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Period: Washout (3 to 14 Days)
Arm/Group | Humalog, Then Humalog + rHuPH20, Then Humulin-R + rHuPH20 | Humalog, Then Humulin-R + rHuPH20, Then Humalog + rHuPH20 | Humalog + rHuPH20, Then Humalog, Then Humulin-R + rHuPH20 | Humalog + rHuPH20, Then Humulin-R + rHuPH20, Then Humalog | Humulin-R + rHuPH20, Then Humalog, Then Humalog + rHuPH20 | Humulin-R + rHuPH20, Then Humalog + rHuPH20, Then Humalog
Started | 3 | 4 | 4 | 4 | 3 | 4
Completed | 3 | 4 | 4 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Humalog, Then Humalog + rHuPH20, Then Humulin-R + rHuPH20 | Humalog, Then Humulin-R + rHuPH20, Then Humalog + rHuPH20 | Humalog + rHuPH20, Then Humalog, Then Humulin-R + rHuPH20 | Humalog + rHuPH20, Then Humulin-R + rHuPH20, Then Humalog | Humulin-R + rHuPH20, Then Humalog, Then Humalog + rHuPH20 | Humulin-R + rHuPH20, Then Humalog + rHuPH20, Then Humalog
Started | 3 | 4 | 4 | 4 | 3 | 4
Completed | 3 | 4 | 4 | 3 | 3 | 4
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Weight loss > 3 kilograms (kg) | 0 | 0 | 0 | 1 | 0 | 0
Period: Washout (3 to 14 Days)
Arm/Group | Humalog, Then Humalog + rHuPH20, Then Humulin-R + rHuPH20 | Humalog, Then Humulin-R + rHuPH20, Then Humalog + rHuPH20 | Humalog + rHuPH20, Then Humalog, Then Humulin-R + rHuPH20 | Humalog + rHuPH20, Then Humulin-R + rHuPH20, Then Humalog | Humulin-R + rHuPH20, Then Humalog, Then Humalog + rHuPH20 | Humulin-R + rHuPH20, Then Humalog + rHuPH20, Then Humalog
Started | 3 | 4 | 4 | 3 | 3 | 4
Completed | 3 | 4 | 4 | 3 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Humalog, Then Humalog + rHuPH20, Then Humulin-R + rHuPH20 | Humalog, Then Humulin-R + rHuPH20, Then Humalog + rHuPH20 | Humalog + rHuPH20, Then Humalog, Then Humulin-R + rHuPH20 | Humalog + rHuPH20, Then Humulin-R + rHuPH20, Then Humalog | Humulin-R + rHuPH20, Then Humalog, Then Humalog + rHuPH20 | Humulin-R + rHuPH20, Then Humalog + rHuPH20, Then Humalog
Started | 3 | 4 | 4 | 3 | 3 | 4
Completed | 3 | 4 | 4 | 3 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received at least 1 dose of Humalog, Humalog + recombinant human hyaluronidase PH20 (rHuPH20), or Humulin-R + rHuPH20 during dose-finding (DV) visits or experimental (data gathering) visits.
Groups:
- Overall Study: Participants who received at least 1 dose of Humalog, Humalog + recombinant human hyaluronidase PH20 (rHuPH20), or Humulin-R + rHuPH20 during dose-finding (DV) visits or experimental (data gathering) visits.
Arm/Group | Overall Study
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: Years (yr)] | 52.2 (8.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 4
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: Participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Postprandial Glucose (PPG) Excursion Following a Liquid Meal
Description: Postprandial glucose (PPG) values in participants receiving Humalog alone, Humalog + recombinant human hyaluronidase PH20 (rHuPH20), or Humulin-R + rHuPH20 following a liquid meal are reported. Blood samples were collected at 30, 20, 10, and within 5 minutes before and at 3, 6, 9, 12, 15, 20, 25, 30, 45, 60, 75, 90, 120, 150, 180, 210, 240, 300, 360, 420, and 480 minutes after injection of each study drug. Least square mean difference was calculated and tested using repeated measures analysis of variance with fixed effect for treatment.
Time Frame: Predose up to 480 minutes after study drug injection
Population: Participants who received at least 1 dose of Humalog alone, Humalog + recombinant human hyaluronidase PH20 (rHuPH20), or Humulin-R + rHuPH20 with evaluable postprandial glucose (PPG) excursion data.
Measure: Least Squares Mean (Standard Deviation); unit: Milligrams per deciliter (mg/dL)
Groups:
- Humalog Alone: Humalog alone: A single, subcutaneous (SC) injection of 0.3- to 0.5-units per kilogram (U/kg) Humalog
- Humalog + rHuPH20: Humalog + rHuPH20: A single, subcutaneous (SC) injection of 0.3- to 0.5-units per kilogram (U/kg) Humalog + 3.75 nanograms per kilogram (ng/kg) recombinant human hyaluronidase PH20 (rHuPH20)
- Humulin-R + rHuPH20: Humulin-R + rHuPH20: A single, subcutaneous (SC) injection of 0.3- to 0.5-units per kilogram (U/kg) Humulin-R + 3.75 nanograms per kilogram (ng/kg) recombinant human hyaluronidase PH20 (rHuPH20)
Arm/Group | Humalog Alone | Humalog + rHuPH20 | Humulin-R + rHuPH20
Number analyzed (Participants) | 21 | 21 | 21
Milligrams per deciliter (mg/dL)
  60-minute PPG | 162.71 (32.28) | 144.67 (28.08) | 169.38 (28.64)
  90-minute PPG | 166.05 (34.53) | 143.62 (30.75) | 166.71 (33.83)
  120-minute PPG | 159.10 (30.73) | 138.24 (32.34) | 159.90 (39.56)
  CBGMax(0-4hr) | 177.81 (33.46) | 165.38 (21.39) | 181.62 (31.61)
Statistical Analysis 1: Comparison: Humalog Alone vs Humalog + rHuPH20; 60 minutes after study drug injection; Test type: Superiority or Other; p = 0.0034, Repeated Measures Analysis of Variance — Treatment comparison of Humalog alone and Humalog + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 2: Comparison: Humalog Alone vs Humulin-R + rHuPH20; 60 minutes after study drug injection; Test type: Superiority or Other; p = 0.2600, Repeated Measures Analysis of Variance — Treatment comparison of Humalog alone and Humulin-R + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 3: Comparison: Humalog + rHuPH20 vs Humulin-R + rHuPH20; 60 minutes after study drug injection; Test type: Superiority or Other; p = 0.0001, Repeated measures Analysis of Variance — Treatment comparison of Humalog + recombinant human hyaluronidase PH20 (rHuPH20) and Humulin-R + rHuPH20
Statistical Analysis 4: Comparison: Humalog Alone vs Humalog + rHuPH20; 90 minutes after study drug injection; Test type: Superiority or Other; p = 0.0039, Repeated Measures Analysis of Variance — Treatment comparison of Humalog alone and Humalog + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 5: Comparison: Humalog Alone vs Humulin-R + rHuPH20; 90 minutes after study drug injection; Test type: Superiority or Other; p = 0.9300, Repeated Measures Analysis of Variance — Treatment comparison of Humalog alone and Humulin-R + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 6: Comparison: Humalog + rHuPH20 vs Humulin-R + rHuPH20; 90 minutes after study drug injection; Test type: Superiority or Other; p = 0.0031, Repeated Measures Analysis of Variance — Treatment comparison of Humalog + recombinant human hyaluronidase PH20 (rHuPH20) and Humulin-R + rHuPH20
Statistical Analysis 7: Comparison: Humalog Alone vs Humalog + rHuPH20; 120 minutes after study drug injection; Test type: Superiority or Other; p = 0.0190, Repeated Measures Analysis of Variance — Treatment comparison of Humalog alone and Humalog + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 8: Comparison: Humalog Alone vs Humulin-R + rHuPH20; 120 minutes after study drug injection; Test type: Superiority or Other; p = 0.9200, Repeated Measures Analysis of Variance — Treatment comparison of Humalog alone and Humulin-R + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 9: Comparison: Humalog + rHuPH20 vs Humulin-R + rHuPH20; 120 minutes after study drug injection; Test type: Superiority or Other; p = 0.0150, Repeated Measures Analysis of Variance — Treatment comparison of Humalog + recombinant human hyaluronidase PH20 (rHuPH20) and Humulin-R + rHuPH20
Statistical Analysis 10: Comparison: Humalog Alone vs Humalog + rHuPH20; Peak postprandial glucose (PPG) values; Test type: Superiority or Other; p = 0.0950, Repeated Measures Analysis of Variance — Treatment comparison of Humalog alone and Humalog + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 11: Comparison: Humalog Alone vs Humulin-R + rHuPH20; Peak postprandial glucose (PPG) values; Test type: Superiority or Other; p = 0.6000, Repeated Measures Analysis of Variance — Treatment comparison of Humalog alone and Humulin-R + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 12: Comparison: Humalog + rHuPH20 vs Humulin-R + rHuPH20; Peak postprandial glucose (PPG) values; Test type: Superiority or Other; p = 0.0310, Repeated Measures Analysis of Variance — Treatment comparison of Humalog + recombinant human hyaluronidase PH20 (rHuPH20) and Humulin-R + rHuPH20

2. Secondary Outcome: Maximum Serum Insulin Concentration (Cmax)
Description: Maximum serum insulin concentration (Cmax) for participants receiving Humalog alone, Humalog + recombinant human hyaluronidase PH20 (rHuPH20), or Humulin-R + rHuPH20 is reported. Blood samples were collected at 30, 20, 10, and within 5 minutes before and at 3, 6, 9, 12, 15, 20, 25, 30, 45, 60, 75, 90, 120, 150, 180, 210, 240, 300, 360, 420, and 480 minutes after injection of each study drug.
Time Frame: Predose up to 480 minutes after study drug injection
Population: Participants who received at least one dose of Humalog alone, Humalog + recombinant human hyaluronidase PH20 (rHuPH20), or Humulin-R + rHuPH20 with evaluable maximum serum insulin concentration (Cmax) data.
Measure: Mean (Standard Deviation); unit: Picomoles per liter (pm/L)
Arm/Group | Humalog Alone | Humalog + rHuPH20 | Humulin-R + rHuPH20
Number analyzed (Participants) | 21 | 21 | 21
Picomoles per liter (pm/L) | 3329.49 (1090.02) | 5661.92 (1307.75) | 3011.56 (962.31)
Statistical Analysis 1: Comparison: Humalog Alone vs Humalog + rHuPH20; Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis of Variance — Treatment comparison of Humalog alone and Humalog + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 2: Comparison: Humalog Alone vs Humulin-R + rHuPH20; Test type: Superiority or Other; p = 0.1800, Repeated Measures Analysis of Variance — Treatment comparison of Humalog alone and Humulin-R + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 3: Comparison: Humalog + rHuPH20 vs Humulin-R + rHuPH20; Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis of Variance — Treatment comparison of Humalog + recombinant human hyaluronidase PH20 (rHuPH20) and Humulin-R + rHuPH20

3. Secondary Outcome: Time To Maximum Serum Insulin Concentration (Tmax)
Description: Time to maximum serum insulin concentration (Tmax) for participants receiving Humalog alone, Humalog + recombinant human hyaluronidase PH20 (rHuPH20), or Humulin-R + rHuPH20 following a liquid meal is reported. Blood samples were collected at 30, 20, 10, and within 5 minutes before and at 3, 6, 9, 12, 15, 20, 25, 30, 45, 60, 75, 90, 120, 150, 180, 210, 240, 300, 360, 420, and 480 minutes after injection of each study drug.
Time Frame: Predose up to 480 minutes after study drug injection
Population: Participants who received at least 1 dose of Humalog alone, Humalog + recombinant human hyaluronidase PH20 (rHuPH20), or Humulin-R + rHuPH20 with evaluable time to maximum serum insulin concentration (Tmax) data.
Measure: Mean (Standard Deviation); unit: Minutes (min)
Arm/Group | Humalog Alone | Humalog + rHuPH20 | Humulin-R + rHuPH20
Number analyzed (Participants) | 21 | 21 | 21
Minutes (min) | 74.29 (36.27) | 43.10 (16.01) | 81.67 (40.26)
Statistical Analysis 1: Comparison: Humalog Alone vs Humalog + rHuPH20; Test type: Superiority or Other; p = 0.0045, Repeated Measures Analysis of Variance — Treatment comparison of Humalog alone and Humalog + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 2: Comparison: Humalog Alone vs Humulin-R + rHuPH20; Test type: Superiority or Other; p = 0.4800, Repeated Measures Analysis of Variance — Treatment comparison of Humalog alone and Humulin-R + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 3: Comparison: Humalog + rHuPH20 vs Humulin-R + rHuPH20; Test type: Superiority or Other; p = 0.0006, Repeated Measures Analysis of Variance — Treatment comparison of Humalog + recombinant human hyaluronidase PH20 (rHuPH20) and Humulin-R + rHuPH20

4. Secondary Outcome: Time to Early 50% Maximum Serum Insulin Concentration (Early[t50%])
Description: Time to early 50% maximum serum insulin concentration (early[t50%]) for participants receiving Humalog alone, Humalog + recombinant human hyaluronidase PH20 (rHuPH20), or Humulin-R + rHuPH20 following a liquid meal is reported. Blood samples were collected at 30, 20, 10, and within 5 minutes before and at 3, 6, 9, 12, 15, 20, 25, 30, 45, 60, 75, 90, and 120 minutes after injection of each study drug.
Time Frame: Predose up to 120 minutes after study drug injection
Population: Participants who received at least 1 dose of Humalog alone, Humalog + recombinant human hyaluronidase PH20 (rHuPH20), or Humulin-R + rHuPH20 with evaluable time to early 50% maximum serum insulin concentration (early[t50%]) data.
Measure: Mean (Standard Deviation); unit: Minutes (min)
Arm/Group | Humalog Alone | Humalog + rHuPH20 | Humulin-R + rHuPH20
Number analyzed (Participants) | 21 | 21 | 21
Minutes (min) | 27.02 (8.67) | 18.71 (5.80) | 21.46 (8.19)
Statistical Analysis 1: Comparison: Humalog Alone vs Humalog + rHuPH20; Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis of Variance — Treatment comparison of Humalog alone and Humalog + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 2: Comparison: Humalog Alone vs Humulin-R + rHuPH20; Test type: Superiority or Other; p = 0.0016, Repeated Measures Analysis of Variance — Treatment comparison of Humalog alone and Humalog + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 3: Comparison: Humalog + rHuPH20 vs Humulin-R + rHuPH20; Test type: Superiority or Other; p = 0.1000, Repeated Measures Analysis of Variance — Treatment comparison of Humalog + recombinant human hyaluronidase PH20 (rHuPH20) and Humulin-R + rHuPH20

5. Secondary Outcome: Time to Late 50% Maximum Serum Insulin Concentration (Late[t50%])
Description: Time to late 50% maximum serum insulin concentration (late[t50%]) for participants receiving Humalog alone, Humalog + recombinant human hyaluronidase PH20 (rHuPH20), or Humulin-R + rHuPH20 following a liquid meal is reported. Blood samples were collected at 30, 20, 10, and within 5 minutes before and at 3, 6, 9, 12, 15, 20, 25, 30, 45, 60, 75, 90, 120, 150, 180, 210, 240, 300, 360, 420, and 480 minutes after injection of each study drug.
Time Frame: Predose up to 480 minutes after study drug injection
Population: Participants who received at least 1 dose of Humalog alone, Humalog + recombinant human hyaluronidase PH20 (rHuPH20), or Humulin-R + rHuPH20 with evaluable time to late 50% maximum serum insulin concentration (late[t50%]) data.
Measure: Mean (Standard Deviation); unit: Minutes (min)
Arm/Group | Humalog Alone | Humalog + rHuPH20 | Humulin-R + rHuPH20
Number analyzed (Participants) | 21 | 21 | 21
Minutes (min) | 206.86 (41.66) | 123.93 (44.59) | 220.33 (51.98)
Statistical Analysis 1: Comparison: Humalog Alone vs Humalog + rHuPH20; Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis of Variance — Treatment comparison of Humalog alone + Humalog + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 2: Comparison: Humalog Alone vs Humulin-R + rHuPH20; Test type: Superiority or Other; p = 0.3000, Repeated Measures Analysis of Variance — Treatment comparison for Humalog alone and Humulin-R + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 3: Comparison: Humalog + rHuPH20 vs Humulin-R + rHuPH20; Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis of Variance — Treatment comparison of Humalog + recombinant human hyaluronidase PH20 (rHuPH20) and Humulin-R + rHuPH20

6. Secondary Outcome: Mean Residence Time From Time 0 to the End of Blood Sampling (MRT[Last])
Description: Mean residence time from time 0 to the end of blood sampling (MRT[last]) for participants who received Humalog alone, Humalog + recombinant human hyaluronidase PH20 (rHuPH20), or Humulin-R + rHuPH20 following a liquid meal is reported. Blood samples were collected at 30, 20, 10, and within 5 minutes before and at 3, 6, 9, 12, 15, 20, 25, 30, 45, 60, 75, 90, 120, 150, 180, 210, 240, 300, 360, 420, and 480 minutes after injection of each study drug.
Time Frame: Predose up to 480 minutes after study drug injection
Population: Participants who received at least 1 dose of Humalog alone, Humalog + recombinant human hyaluronidase PH20 (rHuPH20), or Humulin-R + rHuPH20 with evaluable mean residence time from time 0 to the end of blood sampling (MRT[last]) data.
Measure: Mean (Standard Deviation); unit: Minutes (min)
Arm/Group | Humalog Alone | Humalog + rHuPH20 | Humulin-R + rHuPH20
Number analyzed (Participants) | 21 | 21 | 21
Minutes (min) | 148.79 (22.46) | 108.23 (20.56) | 150.24 (27.32)
Statistical Analysis 1: Comparison: Humalog Alone vs Humalog + rHuPH20; Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis of Variance — Treatment comparison of Humalog alone and Humalog + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 2: Comparison: Humalog Alone vs Humulin-R + rHuPH20; Test type: Superiority or Other; p = 0.7700, Repeated Measures Analysis of Variance — Treatment comparison of Humalog alone and Humulin-R + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 3: Comparison: Humalog + rHuPH20 vs Humulin-R + rHuPH20; Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis of Variance — Treatment comparison of Humalog + recombinant human hyaluronidase PH20 (rHuPH20) and Humulin-R + rHuPH20

7. Secondary Outcome: Area Under the Concentration Time-Curve for Serum Insulin From Time 0 to the End of Blood Sampling (AUC[Last])
Description: Area under the concentration time-curve for serum insulin from time 0 to the end of blood sampling (AUC[last]) for participants who received Humalog alone, Humalog + recombinant human hyaluronidase PH20 (rHuPH20), or Humulin-R + rHuPH20 during a liquid meal is reported. Blood samples were collected at 30, 20, 10, and within 5 minutes before and at 3, 6, 9, 12, 15, 20, 25, 30, 45, 60, 75, 90, 120, 150, 180, 210, 240, 300, 360, 420, and 480 minutes after injection of each study drug. Least squares mean difference was calculated and tested using repeated measures analysis of variance with fixed effect for treatment.
Time Frame: Predose up to 480 minutes after study drug injection
Population: Participants who received at least 1 dose of Humalog alone, Humalog + recombinant human hyaluronidase PH20 (rHuPH20), or Humulin-R + rHuPH20 with evaluable area under the concentration time-curve for serum insulin from time 0 to the end of blood sampling (AUC[last]) data.
Measure: Least Squares Mean (Standard Deviation); unit: Minutes * picomoles /1000 (min*pm/1000)
Arm/Group | Humalog Alone | Humalog + rHuPH20 | Humulin-R + rHuPH20
Number analyzed (Participants) | 21 | 21 | 21
Minutes * picomoles /1000 (min*pm/1000) | 578.67 (144.66) | 668.33 (146.52) | 571.42 (132.04)
Statistical Analysis 1: Comparison: Humalog Alone vs Humalog + rHuPH20; Test type: Superiority or Other; p = 0.0100, Repeated Measures Analysis of Variance — Treatment comparison of Humalog alone and Humalog + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 2: Comparison: Humalog Alone vs Humulin-R + rHuPH20; Test type: Superiority or Other; p = 0.8200, Repeated Measures Analysis of Variance — Treatment comparison of Humalog alone and Humulin-R + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 3: Comparison: Humalog + rHuPH20 vs Humulin-R + rHuPH20; Test type: Superiority or Other; p = 0.0056, Repeated Measures Analysis of Variance — Treatment comparison of Humalog + recombinant human hyaluronidase PH20 (rHuPH20) and Humulin-R + rHuPH20

8. Secondary Outcome: Area Under the Time-Concentration Curve for Blood Glucose (AUC[BG])
Description: Area under the time-concentration curve for blood glucose (AUC[BG]) for participants who received Humalog alone, Humalog + recombinant human hyaluronidase PH20 (rHuPH20), and Humulin-R + rHuPH20 following a liquid meal is reported. AUC(BG) values are reported for participants whose blood glucose (BG) was elevated higher than 160 milligrams per deciliter (mg/dL) or 140 mg/dL, or lower than 70 mg/dL within 4 hours of consuming a liquid meal. Blood samples were collected at 30, 20, 10, and within 5 minutes before and at 3, 6, 9, 12, 15, 20, 25, 30, 45, 60, 75, 90, 120, 150, 180, 210, 240, 300, 360, 420, and 480 minutes after injection of each study drug. Least squares mean difference was calculated and tested using repeated measures analysis of variance with fixed effect for treatment.
Time Frame: Predose up to 480 minutes after study drug injection
Population: Participants who received at least 1 dose of Humalog alone, Humalog + recombinant human hyaluronidase PH20 (rHuPH20), or Humulin-R + rHuPH20 with evaluable area under the time-concentration curve for blood glucose (AUC[BG]) data.
Measure: Least Squares Mean (Standard Deviation); unit: Milligrams per deciliter * minutes
Arm/Group | Humalog Alone | Humalog + rHuPH20 | Humulin-R + rHuPH20
Number analyzed (Participants) | 21 | 21 | 21
Milligrams per deciliter * minutes
  AUC(BG) >160 mg/dL | 2017.46 (2811.82) | 722.82 (1030.52) | 2509.65 (3332.36)
  AUC(BG) >140 mg/dL | 4233.71 (4383.35) | 2696.54 (2548.03) | 4905.92 (4829.71)
  AUC(BG) <70 mg/dL | 571.20 (850.07) | 197.00 (480.75) | 408.50 (602.29)
Statistical Analysis 1: Comparison: Humalog Alone vs Humalog + rHuPH20; Participants with blood glucose (BG) >160 milligrams per deciliter (mg/dL); Test type: Superiority or Other; p = 0.064, Repeated Measures Analysis of Variance — Treatment comparison of Humalog alone and Humalog + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 2: Comparison: Humalog Alone vs Humulin-R + rHuPH20; Participants with blood glucose (BG) >160 milligrams per deciliter (mg/dL); Test type: Superiority or Other; p = 0.47, Repeated Measures Analysis of Variance — Treatment comparison of Humalog alone and Humulin-R + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 3: Comparison: Humalog + rHuPH20 vs Humulin-R + rHuPH20; Participants with blood glucose (BG) >160 milligrams per deciliter (mg/dL); Test type: Superiority or Other; p = 0.012, Repeated Measures Analysis of Variance — Treatment comparison of Humalog + recombinant human hyaluronidase PH20 (rHuPH20) and Humulin-R + rHuPH20
Statistical Analysis 4: Comparison: Humalog Alone vs Humalog + rHuPH20; Participants with blood glucose (BG) >140 milligrams per deciliter (mg/dL); Test type: Superiority or Other; p = 0.099, Repeated Measures Analysis of Variance — Treatment comparison of Humalog alone and Humalog + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 5: Comparison: Humalog Alone vs Humulin-R + rHuPH20; Participants with blood glucose (BG) >140 milligrams per deciliter (mg/dL); Test type: Superiority or Other; p = 0.46, Repeated Measures Analysis of Variance — Treatment comparison of Humalog alone and Humulin-R + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 6: Comparison: Humalog + rHuPH20 vs Humulin-R + rHuPH20; Participants with blood glucose (BG) >140 milligrams per deciliter (mg/dL); Test type: Superiority or Other; p = 0.020, Repeated Measures Analysis of Variance — Treatment comparison of Humalog + recombinant human hyaluronidase PH20 (rHuPH20) and Humulin-R + rHuPH20
Statistical Analysis 7: Comparison: Humalog Alone vs Humalog + rHuPH20; Participants with blood glucose (BG) <70 milligrams per deciliter (mg/dL); Test type: Superiority or Other; p = 0.13, Repeated Measures Analysis of Variance — Treatment comparison of Humalog alone and Humalog + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 8: Comparison: Humalog Alone vs Humulin-R + rHuPH20; Participants with blood glucose (BG) <70 milligrams per deciliter (mg/dL); Test type: Superiority or Other; p = 0.41, Repeated Measures Analysis of Variance — Treatment comparison of Humalog alone and Humulin-R + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 9: Comparison: Humalog + rHuPH20 vs Humulin-R + rHuPH20; Participants with blood glucose (BG) <70 milligrams per deciliter (mg/dL); Test type: Superiority or Other; p = 0.46, Repeated Measures Analysis of Variance — Treatment comparison of Humalog + recombinant human hyaluronidase PH20 (rHuPH20) and Humulin-R + rHuPH20

9. Secondary Outcome: Minimum Postprandial Glucose (PPG)
Description: Minimum postprandial glucose (PPG) in participants who received Humalog alone, Humalog + recombinant human hyaluronidase PH20 (rHuPH20), or Humulin-R + rHuPH20 following a liquid meal is reported. Blood samples were collected at 30, 20, 10, and within 5 minutes before and at 3, 6, 9, 12, 15, 20, 25, 30, 45, 60, 75, 90, 120, 150, 180, 210, 240, 300, 360, 420, and 480 minutes after injection of each study drug.
Time Frame: Predose up to 480 minutes after study drug injection
Population: Participants who received at least 1 dose of Humalog alone, Humalog + recombinant human hyaluronidase PH20 (rHuPH20), or Humulin-R + rHuPH20 with evaluable minimum postprandial glucose (PPG) data.
Measure: Mean (Standard Deviation); unit: Milligrams per deciliter (mg/dL)
Arm/Group | Humalog Alone | Humalog + rHuPH20 | Humulin-R + rHuPH20
Number analyzed (Participants) | 21 | 21 | 21
Milligrams per deciliter (mg/dL) | 76.38 (22.58) | 88.52 (27.37) | 75.62 (20.15)
Statistical Analysis 1: Comparison: Humalog Alone vs Humalog + rHuPH20; Test type: Superiority or Other; p = 0.016, Repeated Measures Analysis of Variance — Treatment comparison of Humalog alone and Humalog + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 2: Comparison: Humalog Alone vs Humulin-R + rHuPH20; Test type: Superiority or Other; p = 0.8800, Repeated Measures Analysis of Variance — Treatment comparison of Humalog alone and Humulin-R + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 3: Comparison: Humalog + rHuPH20 vs Humulin-R + rHuPH20; Test type: Superiority or Other; p = 0.011, Repeated Measures Analysis of Variance — Treatment comparison of Humalog + recombinant human hyaluronidase PH20 (rHuPH20) and Humulin-R + rHuPH20

10. Secondary Outcome: Percentage of Participants Without Hypoglycemia
Description: Percentage of participants who received Humalog alone, Humalog + recombinant human hyaluronidase PH20 (rHuPH20), or Humulin-R + rHuPH20 who did not experience hypoglycemia following a liquid meal is reported. Hypoglycemia was defined as any blood glucose values lower than 70 milligrams per deciliter (mg/dL) or symptoms of hypoglycemia responding to treatment with glucose. Blood samples were collected at 30, 20, 10, and within 5 minutes before and at 3, 6, 9, 12, 15, 20, 25, 30, 45, 60, 75, 90, 120, 150, 180, 210, 240, 300, 360, 420, and 480 minutes after injection of each study drug.
Time Frame: Predose up to 480 minutes after study drug injection
Population: Participants who received at least 1 dose of Humalog alone, Humalog + recombinant human hyaluronidase PH20 (rHuPH20), or Humulin-R + rHuPH20.
Measure: Number; unit: Percentage of participants
Arm/Group | Humalog Alone | Humalog + rHuPH20 | Humulin-R + rHuPH20
Number analyzed (Participants) | 21 | 21 | 21
Percentage of participants | 81.0 | 71.4 | 71.4

11. Secondary Outcome: Time to Percentage of Insulin Exposure (as Measured by Area Under the Curve [AUC])
Description: Time to percentage of exposure to insulin, as measured by area under the curve (AUC), following a liquid meal for participants who received Humalog alone, Humalog + recombinant human hyaluronidase PH20 (rHuPH20), or Humulin-R + rHuPH20 is reported. Blood samples were collected at 30, 20, 10, and within 5 minutes before and at 3, 6, 9, 12, 15, 20, 25, 30, 45, 60, 75, 90, 120, 150, 180, 210, 240, 300, 360, 420, and 480 minutes after injection of each study drug.
Time Frame: Predose up to 480 minutes following after injection of study drug
Population: Participants who received at least 1 dose of Humalog alone, Humalog + recombinant human hyaluronidase PH20 (rHuPH20), or Humulin-R + rHuPH20 with evaluable time to percentage of insulin exposure as measured by area under the curve (AUC) data.
Measure: Mean (Standard Deviation); unit: Minutes (min)
Groups:
- Humulin-R + rHuPH20: Humalog + rHuPH20: A single, subcutaneous (SC) injection of 0.3- to 0.5-units per kilogram (U/kg) Humalog + 3.75 nanograms per kilogram (ng/kg) recombinant human hyaluronidase PH20 (rHuPH20)
Arm/Group | Humalog Alone | Humalog + rHuPH20 | Humulin-R + rHuPH20
Number analyzed (Participants) | 21 | 21 | 21
Minutes (min)
  Time to 10% Insulin Exposure | 46.05 (8.98) | 30.49 (7.13) | 43.41 (10.21)
  Time to 50% Insulin Exposure | 135.73 (21.18) | 94.49 (20.06) | 137.52 (27.35)
Statistical Analysis 1: Comparison: Humalog Alone vs Humalog + rHuPH20; Analysis for 10% of exposure (area under the curve [AUC]); Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis of Variance — Treatment comparison of Humalog alone and Humalog + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 2: Comparison: Humalog Alone vs Humulin-R + rHuPH20; Analysis for 10% of exposure (area under the curve [AUC]); Test type: Superiority or Other; p = 0.1800, Repeated Measures Analysis of Variance — Treatment comparison of Humalog alone and Humulin-R + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 3: Comparison: Humalog + rHuPH20 vs Humulin-R + rHuPH20; Analysis for 10% of exposure (area under the curve [AUC]); Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis of Variance — Treatment comparison of Humalog + recombinant human hyaluronidase PH20 (rHuPH20) and Humulin-R + rHuPH20
Statistical Analysis 4: Comparison: Humalog Alone vs Humalog + rHuPH20; Analysis for 50% of exposure (area under the curve [AUC]); Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis of Variance — Treatment comparison for Humalog alone and Humalog + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 5: Comparison: Humalog Alone vs Humulin-R + rHuPH20; Analysis for 50% of exposure (area under the curve [AUC]); Test type: Superiority or Other; p = 0.7200, Repeated Measures Analysis of Variance — Treatment comparison of Humalog alone and Humulin-R + recombinant human hyaluronidase PH20 (rHuPH20)
Statistical Analysis 6: Comparison: Humalog + rHuPH20 vs Humulin-R + rHuPH20; Analysis for 50% of exposure (area under the curve [AUC]); Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis of Variance — Treatment comparison of Humalog + recombinant human hyaluronidase PH20 (rHuPH20) and Humulin-R + rHuPH20

ADVERSE EVENTS:
Description: Adverse events were classified by the body system affected.
Groups:
- Humalog Alone: Participants who received a subcutaneous (SC) injection of 0.3- to 0.5-units per kilogram (U/kg) of Humalog alone for up to 3 dose-finding (DF) visits (each visit separated by a 3- to 14-day washout period), followed by a SC injection of the appropriate dose of Humalog during Periods 1, 2, or 3 of the study.
- Humalog + rHuPH20: Participants who received a subcutaneous (SC) injection of 0.3- to 0.5-units per kilogram (U/kg) of Humalog + 3.75 nanograms per kilogram (ng/kg) recombinant human hyaluronidase PH20 (rHuPH20) for up to 3 dose-finding (DF) visits (each visit separated by a 3- to 14-day washout), followed by a single SC injection of the appropriate dose of Humalog + rHuPH20 during Periods 1, 2, or 3 of the study.
- Humulin-R + rHuPH20: Participants who received a subcutaneous (SC) injection of 0.3- to 0.5-units per kilogram (U/kg) of Humulin-R + 3.75 nanograms per kilogram (ng/kg) of recombinant human hyaluronidase PH20 (rHuPH20) for up to 3 dose-finding (DF) visits (each visit separated by a 3- to 14-day washout), followed by a single SC injection of the appropriate dose of Humulin-R + rHuPH20 during Periods 1, 2, or 3 of the Study
Arm/Group | Humalog Alone | Humalog + rHuPH20 | Humulin-R + rHuPH20
Serious Adverse Events (participants affected / at risk) | 0/22 | 1/22 | 0/22
Other Adverse Events (participants affected / at risk) | 11/22 | 5/22 | 10/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Humalog Alone (N=22) | Humalog + rHuPH20 (N=22) | Humulin-R + rHuPH20 (N=22)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Humalog Alone (N=22) | Humalog + rHuPH20 (N=22) | Humulin-R + rHuPH20 (N=22)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 0 (0) | 2 (4)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Induration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Nodule on extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days